CLINICAL TRIAL: NCT00013065
Title: A Medication Adherence Intervention for HIV Infected Veterans
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: HII 99-054
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-01

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
It is estimated that the VHA is caring for nearly 40 percent of all HIV-infected veterans. To benefit from recent improvements in anti-HIV therapy, patients need to take their medications consistently.

DETAILED DESCRIPTION:
Background:

It is estimated that the VHA is caring for nearly 40 percent of all HIV-infected veterans. To benefit from recent improvements in anti-HIV therapy, patients need to take their medications consistently.

Objectives:

Optimizing health for HIV patients requires excellent adherence to antiretroviral medication regimens. However, its unclear how best to incorporate adherence education and support programs into VA HIV outpatient care. We implemented and evaluated a pharmacist program (ACE) and a Pager reminder program to support adherence in veterans with HIV.

Methods:

We used a quasi-experimental design with pre-post evaluation at four VA Centers. Three treatment conditions (ACE, Pager, Usual Care) were rolled-in sequentially over two study phases, allowing for group comparisons between conditions. ACE is a multi-component manualized 4-session, individual patient education and support program by trained pharmacists. The Pager intervention used alphanumeric pagers to remind patients of dosing times. Electronically-monitored medication adherence (MEMS), self-report questionnaires, and pharmacy refill records were collected. Qualitative site interviews were collected before and after interventions to assist with program evaluation. Multilevel mixed models were used to analyze main study outcomes over time. Secondary analyses compared subgroup who actually received all ACE sessions (�as treated�) to controls.

Status:

Project has been completed and Final Report submitted to HSR&D CO.

ELIGIBILITY:
Inclusion Criteria:

Patients must be greater than or equal to 18 years old, must be enrolled in HIV Primary care at one of 4 VA study sites and be taking antiretroviral therapy.

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen L. Gifford, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (4):
- United States (4):
  - Southern Arizona VA Health Care System, Tucson, AZ, Tucson, Arizona
  - VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California

REFERENCES:
- [Result] Shively M, Smith TL, Bormann J, Gifford A. Evaluating Self-Efficacy for HIV Disease Management Skills. AIDS and behavior. 2002 Dec 1; 6(4):371-379.
- [Result] Gifford AL, Groessl EJ. Chronic disease self-management and adherence to HIV medications. J Acquir Immune Defic Syndr. 2002 Dec 15;31 Suppl 3:S163-6. doi: 10.1097/00126334-200212153-00016. PMID 12562043
- [Result] Gifford AL, Bormann JE, Shively MJ, Wright BC, Richman DD, Bozzette SA. Predictors of self-reported adherence and plasma HIV concentrations in patients on multidrug antiretroviral regimens. J Acquir Immune Defic Syndr. 2000 Apr 15;23(5):386-95. doi: 10.1097/00126334-200004150-00005. PMID 10866231
- [Result] Korthuis PT, Asch S, Mancewicz M, Shapiro MF, Mathews WC, Cunningham WE, McCutchan JA, Gifford A, Lee ML, Bozzette SA. Measuring medication: do interviews agree with medical record and pharmacy data? Med Care. 2002 Dec;40(12):1270-82. doi: 10.1097/01.MLR.0000036410.86742.27. PMID 12458308
- [Result] Bormann J, Shively M, Smith TL, Gifford AL. Measurement of fatigue in HIV-positive adults: reliability and validity of the Global Fatigue Index. J Assoc Nurses AIDS Care. 2001 May-Jun;12(3):75-83. doi: 10.1016/S1055-3290(06)60146-5. PMID 11387807